CLINICAL TRIAL: NCT03180502
Title: A Phase II Randomized Trial of Proton Vs. Photon Therapy (IMRT) for Cognitive Preservation in Patients With IDH Mutant, Low to Intermediate Grade Gliomas
Brief Title: Proton Beam or Intensity-Modulated Radiation Therapy in Preserving Brain Function in Patients With IDH Mutant Grade II or III Glioma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NRG-BN005; NCI-2017-00203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN005; NRG-BN005 (Other: NRG Oncology); NRG-BN005 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligoastrocytoma; Anaplastic Oligodendroglioma; Diffuse Astrocytoma; Glioma; Oligoastrocytoma; Oligodendroglioma; WHO Grade 3 Glioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioma | interventions — Specimen Handling; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Proton Therapy; Protons; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (photon-based IMRT, temozolomide) (Active Comparator): Patients undergo photon-based IMRT QD, 5 days a week for 6 weeks for a total of 30 fractions. Beginning 28 days after completion of radiation therapy, patients receive standard of care temozolomide for 5 days. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression of unacceptable toxicity. Patients undergo MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide
- Arm II (proton beam radiation therapy, temozolomide) (Experimental): Patients undergo proton beam radiation therapy QD, 5 days a week for 6 weeks for a total of 30 fractions. Beginning 28 days after completion of radiation therapy, patients receive standard of care temozolomide for 5 days. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression of unacceptable toxicity. Patients undergo MRI and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Procedure: Magnetic Resonance Imaging; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm I (photon-based IMRT, temozolomide)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Radiation: Proton Beam Radiation Therapy — Undergo proton beam radiation therapy
  Other Names: External beam radiation therapy protons (procedure); External Beam Radiotherapy (protons); PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; PROTON Therapy; Radiation, Proton Beam
  Arms: Arm II (proton beam radiation therapy, temozolomide)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Temozolomide — Drug
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This randomized phase II clinical trial studies the side effects and how well proton beam or intensity-modulated radiation therapy works in preserving brain function in patients with IDH mutant grade II or III glioma. Proton beam radiation therapy uses tiny charged particles to deliver radiation directly to the tumor and may cause less damage to normal tissue. Intensity-modulated or photon beam radiation therapy uses high-energy x-ray beams shaped to treat the tumor and may also cause less damage to normal tissue. It is not yet known if proton beam radiation therapy is more effective than photon-based beam intensity-modulated radiation therapy in treating patients with glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether proton therapy, compared to intensity-modulated radiation therapy (IMRT), preserves cognitive outcomes over time as measured by the Clinical Trial Battery Composite (CTB COMP) score (calculated from the Hopkins Verbal Learning Test Revised [HVLT-R]) Total Recall, HVLT-R Delayed Recall, HVLT-R Delayed Recognition, Controlled Oral Word Association (COWA) test, Trail Making Test (TMT) part A and part B.

SECONDARY OBJECTIVES:

I. To assess whether treatment with proton therapy preserves neurocognitive function as measured separately by each test, HVLT-R, TMT parts A & B, and COWA.

II. To document and compare treatment related symptoms, overall symptom impact, and disease related factor groupings, utilizing the M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT), for both treatment arms.

III. To assess whether treatment with proton therapy, compared to IMRT, results in superior quality of life as measured by the Linear Analog Scale Assessment (LASA) scale.

IV. To compare local control patterns of failure and overall and progression-free survival between the two treatment arms.

V. To assess adverse events. VI. To compare Illumnia MethylationEPIC beadchip array-derived IDH and 1p19q status determined centrally to that submitted by enrolling sites.

TERTIARY OBJECTIVES:

I. To assess the impact of chemotherapy use on cognitive outcomes, symptom outcomes and quality of life.

II. To assess dose-response relationships between neuro-anatomic dosimetry and cognitive outcomes within and between treatment arms.

III. To evaluate the association between tumor molecular status and cognition at baseline and within and between treatment arms over time.

IV. To assess patterns of failure and pseudo progression as a function of radiation delivery type and dose received.

V. To assess local control, overall survival and, progression free survival in IDH mutant grade II and III tumors.

VI. To collect blood samples for future studies seeking to correlate changes in peripheral blood biomarkers (genes, micro ribonucleic acid [RNA], proteins, lymphocyte count, melatonin, etc) and the study endpoints.

VII. To document and compare the impact of low to intermediate gliomas and therapy on patients' work and activity participation (The Work Productivity and Activity Impairment [WPAI:GH] Questionnaire: General Health version 2.0) as well as the relationship between changes in patients' work and activity participation and neurocognitive function and patient reported symptoms and interference.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo photon-based IMRT once daily (QD), 5 days a week for 6 weeks for a total of 30 fractions. Beginning 28 days after completion of radiation therapy, patients receive standard of care temozolomide for 5 days. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression of unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI) and collection of blood samples throughout the trial.

ARM II: Patients undergo proton beam radiation therapy QD, 5 days a week for 6 weeks for a total of 30 fractions. Beginning 28 days after completion of radiation therapy, patients receive standard of care temozolomide for 5 days. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression of unacceptable toxicity. Patients undergo MRI and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 6 and 12 months and then yearly for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* Tumor tissue must be available for submission for central pathology review
* Grade II and III gliomas IDH mutant gliomas including; diffuse astrocytoma, anaplastic astrocytoma, oligodendroglioma, anaplastic oligodendroglioma, oligoastrocytoma, anaplastic oligoastrocytoma
* Documentation from the enrolling site confirming the presence of IDH mutation and 1p/19q status; the provided information must document assays performed in clinical laboratory improvement amendments (CLIA)-approved laboratories and be uploaded prior to Step 2 registration
* Age >= 18
* The trial is open to both genders
* Only English or French speaking patients are eligible to participate as the cognitive assessments are only available in these languages
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* History and physical exam, and Karnofsky performance status of >= 70 within 30 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (within 60 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 60 days prior to registration)
* Hemoglobin >= 10.0 g/dl (Note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable) (within 60 days prior to registration)
* Bilirubin =< 1.5 upper limit of normal (ULN) (within 60 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 60 days prior to registration)
* Blood urea nitrogen (BUN) < 30 mg/dl (within 60 days prior to registration)
* Serum creatinine < 1.5 mg/dl (within 60 days prior to registration)
* Pre-operative MRI imaging of the brain available for radiation planning
* Post-operative MRI imaging with contrast is mandatory obtained for radiation therapy planning; enrolling sites are not mandated although highly encouraged to obtain thin-slice (< 1.5 mm) 3 dimensional (D) pre and post contrast and axial T2/FLAIR sequences for planning purposes
* Patients must be able to swallow capsules
* PRIOR TO STEP 2 REGISTRATION
* Histologically proven diagnosis of supratentorial, World Health Organization (WHO) grade II or III astrocytoma, oligodendroglioma or oligoastrocytoma, with IDH mutation confirmed by central review
* The following baseline neurocognitive assessments must be completed and uploaded prior to Step 2 registration: HVLT-R (recall, delayed recall, and recognition), TMT Parts A and B, and COWA; the neurocognitive assessment will be uploaded into a folder in the NRG Medidata RAVE System for central evaluation; once the upload and scoring of the tools are complete, a notification will be sent within 3 business days to the Research Associate (RA) to proceed to Step 2; in order for the patient to be eligible, at least 5 of the 6 neurocognitive assessments must be able to be scored (i.e. free of any errors)
* Completion of all items on the following baseline quality of life forms: MDASI-BT, LASA QOL, WPAI-GH and Employment Questionnaire; these quality of life forms will be required and data entered at step 2 registration
* Financial clearance for proton therapy treatment prior step 2 registration
* Women of childbearing age must have a negative serum pregnancy test within 14 days prior to step 2 registration

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease; if applicable
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years; (for example, carcinoma in situ of the breast, oral cavity or cervix are permissible)
* Prior cranial radiotherapy or radiotherapy to the head and neck where potential field overlaps would exist
* Prior chemotherapy or radiotherapy for any brain tumor
* Histologic diagnosis of glioblastoma (WHO grade IV) or pilocytic astrocytoma (WHO grade I)
* Definitive evidence of multifocal disease
* Planned use of cytotoxic chemotherapy during radiation (only adjuvant temozolomide therapy will be used on this protocol)
* Patients with infra-tentorial tumors are not eligible
* Prior history of neurologic or psychiatric disease believed to impact cognitive function
* The use of memantine during or following radiation is NOT allowed
* Severe, active co-morbidity defined as follows:

  * Unstable angina or congestive heart failure requiring hospitalization within 6 months prior to enrollment
  * Transmural myocardial infarction within the last 6 months prior to registration; evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 28 days prior to registration (Note: EKG to be performed only if clinical suspicion of cardiac issue)
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to registration
  * Serious and inadequately controlled arrhythmia at step 2 registration
  * Serious or non-healing wound, ulcer or bone fracture or history of abdominal fistula, intra-abdominal abscess requiring major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to registration, with the exception of the craniotomy for surgical resection
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Human immunodeficiency virus (HIV) positive with CD4 count < 200 cells/microliter; acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that HIV testing is not required for entry into this protocol
  * Any other severe immunocompromised condition
  * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
  * End-stage renal disease (i.e., on dialysis or dialysis has been recommended)
  * Any other major medical illnesses or psychiatric treatments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Inability to undergo MRI with and without contrast (e.g. claustrophobia, non-MRI compatible implant or foreign body, gadolinium allergy or renal dysfunction preventing the patient from receiving gadolinium- institutional guidelines should be used to determine if patients are at risk for renal dysfunction); note that patients with severe claustrophobia are permitted on this study if they are willing and able to undergo MRI with adequate sedation or anesthesia
* Patients known to have hypersensitivity to dacarbazine (DTIC) are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in cognition as measured by the Clinical Trial Battery Composite (CTB COMP) score | Baseline to up to 10 years
  Assessed with a general linear model with maximum likelihood estimation. Three models will be conducted. Baseline CTB COMP score, treatment arm, time, treatment by time interaction (if significant) and stratification factors will be included in the model for the primary endpoint. A second model will be built with these same variables and relevant covariates, such as total volume of intracranial disease, gross tumor volume (GTV) and clinical tumor volume (CTV) size, histology, anti-epileptic use, and disease response to therapy (as measured by Response Assessment in Neuro-Oncology [RANO] criteria). Other than baseline score CTB COMP, treatment arm, and time, only covariates with a p-value < 0.10 will be retained in the model. A third model will be conducted at 10 years using the additional time points of neurocognitive assessments.

SECONDARY OUTCOMES:
Cognition as measured individually by Hopkins Verbal Learning Test Revised (HVLT-R), Trail Making Test (TMT) parts A and B, and Controlled Oral Word Association (COWA) | Up to 10 years
  The HVLT-R, TMT parts A & B, and COWA will be analyzed independently using a general linear model with maximum likelihood estimation. Standardized scores will be used.
Change in symptoms as measured by M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT) | Baseline to up to 10 years
  The change from baseline to each follow-up time point (calculated as baseline score subtracted from follow-up score) will be compared between treatment arms using a t-test, or Wilcoxon test if the data is not normally distributed. A reduced one-sided significance level will be used for the multiple comparisons in the MDASI-BT using the Bonferroni adjustment (alpha=0.017 for disease related factors and alpha=0.025 for treatment related symptoms and overall impact). A general linear model with maximum likelihood estimation will be used to assess symptom trends across time. Baseline score, treatment arm, time, treatment by time interaction (if significant), stratification factors, and relevant covariates, such as total volume of, GTV and CTV size, histology, anti-epileptic use, and disease response to therapy (as measured by RANO criteria) will be included as covariates in each model.
Change in quality of life as measured by the Linear Analog Scale Assessment (LASA) scale | Up to 10 years
  The change from baseline to each follow-up time point (calculated as baseline score subtracted from follow-up score) will be compared between treatment arms using a t-test, or Wilcoxon test if the data is not normally distributed. A one-sided alpha=0.05 will be used for the LASA. A general linear model with maximum likelihood estimation will be used to assess symptom and QOL trends across time. Baseline score, treatment arm, time, treatment by time interaction (if significant), stratification factors, and relevant covariates, such as total volume of, GTV and CTV size, histology, anti-epileptic use, and disease response to therapy (as measured by RANO criteria) will be included as covariates in each model. Other than baseline score, treatment arm, and time, only covariates with a p-value < 0.10 will be retained in the model.
Overall survival (OS) | From randomization to the date of death, assessed up to 10 years
  OS will be estimated using the Kaplan-Meier method and compared between arms using the log rank test. Cox proportional hazards models will be used for OS adjusting for treatment arm and stratification factors.
Local control as assessed by Response Assessment in Neuro-Oncology (RANO) criteria | Up to 10 years
  Local control will be estimated using cumulative incidence, treating death prior to an event as a competing risk. Gray's test will be used to compare local control rates between arms. Cause-specific Cox proportional hazards models will be used for local control, adjusting for treatment arm and stratification factors. A two-sided significance level of 0.05 will be used for comparisons between arms.
Progression-free survival (PFS) | From date of randomization to date of progression or death, whichever occurs first, assessed up to 10 years
  A confidence interval will be used to determine if the PFS rate in the proton arm is greater than that in the photon at 1 year. PFS will be estimated using the Kaplan-Meier method and compared between arms using the log rank test. Cox proportional hazards models will be used for PFS adjusting for treatment arm and stratification factors.
Incidence of adverse events (AEs) graded according to the National Cancer Institute's Common Terminology for Adverse Events version 5.0 | Up to 10 years
  Counts of all AEs by grade will be provided by treatment arm. Counts and frequencies will be provided for the worst grade AE experienced by the patient by treatment arm. Grade 3+ treatment related AEs will be compared between arms using a chi-square test, or Fisher's exact test if cell frequencies are < 5, at the one-sided 0.05 significance level.
IDH mutation as assessed by sequencing and 1p19q status as assessed by fluorescence in situ hybridization | Baseline
  A single test will be done for both IDH and 1p19q testing centrally while sites will perform a separate test for IDH and 1p19q. The results from the central and site testing will be compared using the kappa statistic. The asymptotic test of H0: k=0 will be performed using the Z-statistic to determine the strength of agreement. Concordance and discordance rates will be tabulated.

OTHER OUTCOMES:
Impact of chemotherapy use on cognition assessed by Clinical Trial Battery Composite (CTB COMP) and each individual test score | Up to 10 years
  Cognition will be compared between patients who have completed chemotherapy per protocol and those who have not.
Assessment of dose-response relationships | Up to 10 years
  The dose-response relationship between cognition, using the CTB COMP and each individual test score, and neuro-anatomic dosimetry, including the hippocampus and whole brain, will be assessed. The decline, as calculated using the Reliable Change Index, will be used to determine neurocognitive impairment. The dose-response curve will be modeled using a non-linear model.
Assessment of tumor molecular status | Up to 10 years
  Cognition, using the CTB COMP and each individual test score, will be compared by 1p19q status. A general linear model using maximum likelihood estimation will be built for CTB COMP and each individual test score over time including baseline test score, 1p19q status, treatment arm, and stratification factors.
Assessment of patterns of failure and pseudoprogression as a function of radiation delivery type | Up to 10 years
  Cox models will also be built to assess the effect of radiation delivery type on patterns of failure while adjusting for stratification factors. Patterns of failure refer to local failure (within high dose), marginal failure (at edge of treatment field) or distant failure (outside radiation volume). The association of pseudoprogression, a yes/no variable, and radiation delivery type at each follow-up time point will be assessed using a Chi-square test or Fisher's exact test if the cell size is < 5. Pseudoprogression by treatment arm at each follow-up time point will also be assessed using a Chi-square test or Fisher's exact test if the cell size is < 5.
Work and activity participation as measured by the Work Productivity and Activity Impairment Questionnaire: General Health version 2.0 (WPAI:GH) | Up to 2 years
  The distributions of each item and outcome measure of the WPAI will be tabulated at each time point. The association between each of the four WPAI outcomes and NCF, as measured by the CTB COMP score and each NCF test separately, and symptoms, as measured by the MDASI-BT total symptom burden score and total interference score, will be assessed using Pearson correlation coefficients at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: David R Grosshans, Principal Investigator — NRG Oncology
Locations (34):
- United States (34):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Miami Cancer Institute, Miami, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington